CLINICAL TRIAL: NCT04034199
Title: Efficacy of Denosumab and Zoledronic Acid in the Treatment of Idiopathic Inflammatory Myopathies Related Reduced Bone Mineral Density: a Prospective Controlled Trial
Brief Title: Treating Idiopathic Inflammatory Myopathies Related Reduced Bone Mineral Density With Denosumab or Zoledronic Acid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kwong Wah Hospital (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Tang Yan Ki, Principal investigator, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kwh_rheumat_tyk_01
Record Dates: First submitted 2019-07-04; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Inflammatory Myopathies; Osteoporosis, Osteopenia
Keywords: denosumab; zoledronic acid
MeSH Terms: conditions — Myositis; Osteoporosis; Bone Diseases, Metabolic | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: This is a prospective open-label controlled trial. All patients will continue calcium (1000mg daily) and vitamin D supplementation (at least 800 international unit daily). Patients with osteopenia or osteoporosis in a baseline DEXA scan will be randomized by computer-generated blocks in 1:1 ratio into receiving denosumab (treatment group) or zoledronic acid (controlled group). Denosumab is given at 60mg subcutaneously every 6 months, following the FDA approved dosage. Zoledronic acid is administered intravenously at 5mg yearly. DEXA scan will be repeated after 12 months of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab group (Experimental): Patients randomized into the denosumab group will receive denosumab 60mg subcutaneously every 6 months, for a total duration of 1 year. DEXA scan would be repeated at 1 year.
  Interventions: Drug: Denosumab
- Zoledronic acid (Active Comparator): Patients randomized into the denosumab group will receive one dose of zoledronic acid at 5mg intravenously. DEXA scan would be repeated at 1 year.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Denosumab — Denosumab is a human monoclonal antibody against receptor activator of nuclear factor kappa-B ligand (RANKL) and its use is associated with a reduced risk of vertebral, non-vertebral and hip fracture in post-menopausal women. RANKL plays a crucial role in the pathogenesis of glucocorticoid-induced osteoporosis (GIOP). Its production is increased by GC, resulting in stimulated osteoprotegerin ligand production and increased bone resorption. Recent randomized controlled trial from Saag et al have shown that denosumab is more efficacious than risedronate in the improvement of BMD in GIOP patients. Denosumab has been confirmed efficacious in GIOP patients but its efficacy in high-risk osteopenia patients are not well studied. It is given subcutaneously at 60mg every 6 months.
  Other Names: Prolia
  Arms: Denosumab group
Drug: Zoledronic Acid — Zoledronic acid belongs to bisphosphonates and is licensed for the treatment of GIOP and 2 RCTs found zoledronic acid has superior efficacy in improvement in BMD at lumbar spine or femoral neck at 12 months when compared to risedronate. It is given intravenously every year at a dosage of 5mg.
  Other Names: Aclasta
  Arms: Zoledronic acid

SUMMARY:
Idiopathic inflammatory myopathies (IIM) patients are at high risk of development of reduced bone mineral density due to impairment of functional status due to the disease and a relatively high dose of glucocorticoid use for the treatment. Reduced bone mineral density is prevalent in local IIMs patients. Denosumab and zoledronic acid are established treatments for osteoporosis in postmenopausal women and glucocorticoid-induced osteoporosis. However, the role of these treatments in reduced bone mineral density including osteoporosis and osteopenia related to IIMs are lacking. There is also no evidence on comparing the efficacy of the two agents. Therefore, the investigators conducted this prospective randomized controlled study to compare the efficacies of denosumab and zoledronic acid in treating reduced bone mineral density in IIMs patients. The hypothesis in this study is that treatment by denosumab or zoledronic acid would improve bone mineral density in IIMs patients with reduced bone mineral density.

DETAILED DESCRIPTION:
Background:

With recent advances in diagnoses and classification of idiopathic inflammatory myopathies (IIM), an increasing number of newly diagnosed cases of IIM is expected. These patients are vulnerable to the development of Glucocorticoid-induced osteoporosis (GIOP) due to impaired mobility related to musculoskeletal involvement and the relatively high doses of glucocorticoid (GC) required for disease control. Reduced bone mineral density is prevalent among IIM patients shown in the previous local study: osteoporosis and osteopenia are seen in 23.7% and 47.4% of IIM patients respectively. 10% of patients on long term GC treatment sustain a fracture and up to 30-40% of patients are found to have radiological vertebral fractures. Compared to GIOP, the treatment for patients with osteopenia is less well addressed in current guidelines for the management of GIOP. Treatment is usually indicated in patients with a previous history of prior low energy fracture and high fracture risks determined by FRAX score. However, IIMs remain a rare disease entity and IIMs patients are at particularly high risk for osteoporosis and its complications due to a relatively high dose of steroid use and functional impairment from the disease. Therefore, traditional fracture risks assessment tool might not be able to fully assess the fracture risks in this subgroup of patients.

Denosumab is a human monoclonal antibody against receptor activator of nuclear factor kappa-B ligand (RANKL) and its use is associated with a reduced risk of vertebral, non-vertebral and hip fracture in post-menopausal women. A recent randomized controlled trial has shown that denosumab is more efficacious than risedronate in the improvement of BMD in GIOP patients. Denosumab has been confirmed efficacious in GIOP patients but its efficacy in high-risk osteopenia patients are not well studied. On the other hand, zoledronic acid is licensed for the treatment of GIOP and trials found zoledronic acid improve bone mineral density at the lumbar spine or femoral neck at 12 months of treatment. Current evidence comparing the efficacy between denosumab and zoledronic acid is lacking.

In this prospective study, the investigators aimed to assess the efficacy of denosumab and zoledronic acid in the treatment of IIMs patients with reduced bone mineral density.

Study methods This is a prospective open-label controlled trial. All IIMs patients followed up in Kwong Wah Hospital are invited to participate in this study. Eligibility, inclusion, and exclusion criteria are described in details in subsequent sessions. All included patients will have dual-energy X-Ray absorptiometry (DEXA) scan performed at baseline. All participants will continue calcium (1000mg daily) and vitamin D supplementation (at least 800 international unit daily). Patients with osteopenia or osteoporosis in a baseline DEXA scan will be randomized by computer-generated blocks in 1:1 ratio into receiving denosumab (treatment group) or zoledronic acid (controlled group). Denosumab is given at 60mg subcutaneously every 6 months, following the FDA approved dosage. Zoledronic acid is administered intravenously at 5mg yearly. DEXA scan will be repeated after 12 months of treatment.

All participants will be interviewed and examined at the time of recruitment and at subsequent follow-up visits. Patients enrolled in the study will attend follow-up visits at least every 4 months with monitoring of adverse events associated with denosumab or zoledronic acid use. In case of severe adverse events, treatment will be terminated, and patients will be withdrawn from this study.

Demographic data including age, sex, ethnicity, body weight and height, menopausal status, parity, smoking and drinking history, and comorbidities will be recorded. Diagnosis and classification of IIM according to Bohan and Peter criteria (14) and duration of the disease will also be documented. Details of treatment regime including dosage of GCs at time of recruitment, cumulative GCs dosage, concomitant immunosuppressants, and medication history will be recorded. Personal history of previous vertebral or osteoporotic fracture and avascular necrosis will be screened. Complications related to IIMs which included interstitial lung disease, dysphagia and malignancy and Health assessment questionnaire disability index (HAQ-DI) at baseline will be documented. Blood results including serum albumin level, C reactive protein (CRP), erythrocyte sedimentation rate (ESR) and creatine kinase (CPK) will be measured at baseline and upon follow-up visits.

BMD results are recorded in terms of absolute value, T-score (Number of standard deviations above or below mean results of young adults) and Z-score (Number of standard deviations above or below mean results of the age-matched population). Radiographs of the thoracic and lumbar spine will be performed at enrolment and at the completion of the study to look for vertebral collapses. Vertebral collapse is defined as a loss of at least 25% height of vertebrae. Fractures and new vertebral collapse during the study period will be documented.

IIMs disease activity at baseline is measured by physician's and patient's global assessment by visual analog scale, manual muscle testing 8 (MMT8) and Myositis Disease Activity Assessment Visual Analogue Scale (MYOACT).

BMD at the lumbar spine (L1-4), hip and femoral neck are measured by DEXA scan using Hologic Discovery DXA system (Model: Discovery W, Hologic, Bedford, USA) The reference ranges for T-score for Male and Female are derived from a database from the University of Hong Kong, using matched Hong Kong Male and female data. The technicians responsible for reading DEXA images are blinded for the details of the study.

Patients are invited to join this study from August June 2019 to December 2019. Baseline DEXA scan and randomization will be performed within 1 month of study enrolment. Participants would receive 12 months of treatment and DEXA scan will be repeated within 1 month upon completion of treatment. The study and subsequent analyses will be completed by March 2021.

For the estimation in sample size, the mean baseline BMD in GIOP patients from local data is 0.87 g/cm2 with a standard deviation of 0.085 g/cm2. The expected increase in BMD after 12 months of denosumab treatment is 8% compared to placebo whereas zoledronic acid is associated with a 6-7% increase in BMD when compared to placebo. Sample size calculated is 23 patients in each group assuming 5% type I error and 80% power.

For statistical analysis, descriptive statistics for demographic and clinical data are expressed as mean +/- standard deviation if they are normally distributed or as median and range otherwise. Independent Student's t-test is used for analyzing continuous variables with normal distribution and Chi-square test for categorical variables. Differences in BMD between the two groups is compared with paired t-test. After adjustment of confounding factor, analysis of covariance method (general linear model) will be done. Covariates adjusted include age, sex, BMI, smoking and drinking status, duration of menopause in female patients, duration of GC and cumulative dosage of GC. For assessing risk factors associated with reduced BMD, associations between the continuous variables and BMD is assessed by Pearson's correlation test. Univariate analysis followed by multiple linear regression model is used to identify the independent variables for BMD. A P-value of < 0.05 is considered as statistically significant. SPSS 25 will be used for statistical analysis.

This study is approved by the local ethical committee - Research Ethics Application (Kowloon Central/Kowloon East) and is conducted in full accordance with the Helsinki Declaration. Written consent is obtained from all participants. Serious adverse events will be reported to the research and ethics committee.

This is an investigator-initiated study not supported by any pharmaceutical company. The authors have no conflicts of interest to declare.

Outcome measures will be described in subsequent sessions.

ELIGIBILITY:
All idiopathic inflammatory myopathies (IIMs) patients under follow-up in Kwong Wah Hospital are invited to participate in this study.

IIMs are diagnosed by rheumatologist according to Bohan and Peter Criteria. Eligible patients will have dual-energy X-ray absorptiometry (DEXA) scan performed at baseline.

Inclusion Criteria:

1. Adult patients of at least 18 years of age and
2. Evidence of reduced BMD in osteopenia (defined by T-score of -0.1 to -2.5) or osteoporosis range (defined by T-score of < -2.5) at baseline by dual-energy X-ray absorptiometry (DEXA) scan.

Exclusion Criteria:

1. Pregnant patients
2. Patients with juvenile onset of disease (<18 years of age)
3. Patients with pre-existing metabolic bone conditions
4. Patients who are already on osteoporotic treatment other than calcium and vitamin D (including bisphosphonates, denosumab, teriparatide, raloxifene or strontium)
5. Patients who are contraindicated to denosumab or zoledronic acid including severe renal impairment and hypersensitivity
6. Patients who are not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density at 12 months in denosumab and zoledronic acid group | 12 months
  The primary outcome is change in bone mineral density at lumbar spine and hip measured by DEXA between the denosumab and zoledronic acid groups compared to control group at 12 months. Differences in BMD between two groups is compared with paired t-test.

SECONDARY OUTCOMES:
Prevalence of osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Prevalence of osteoporosis and osteopenia in idiopathic inflammatory myopathies patients at baseline. Osteoporosis is defined by a T score of <-2.5 on DEXA scan and osteopenia is defined by T score between -1.0 and -2.5 by DEXA scan.
Comparison of Change in Bone Mineral Density at lumbar spine and hip between the two treatment groups (denosumab and zoledronic acid) | 12 months
  Comparison of Change in Bone mineral density at lumbar spine and hip between the two treatment groups (denosumab and zoledronic acid), as measured by Dual energy X-ray absorptiometry (DEXA scan). Differences in BMD between two groups is compared with paired t-test.
Gender as a risk factor for osteoporosis and osteopenia in IIMs patients | at baseline
  Gender of participants would be recorded. Chi-square test will be used to compare categorical variables.
Smoking status as a risk factor for osteoporosis and osteopenia in IIMs patients | at baseline
  Smoking status (Never smoker, ex-smoker and current smoker) of the participantss would be recorded. Chi-square test will be used to compare categorical variables.
Drinking status as a risk factor for osteoporosis and osteopenia in IIMs patients | at baseline
  Drinking status (Nondrinker, Social drinker, ex-drinker and current drinker) of the participantss would be recorded. Units of alcohol comsumption per week would be recorded.
Menopausal status as a risk factor for osteoporosis and osteopenia in IIMs patients | at baseline
  In female patients, menopausal status (pre-menopausal and menopausal) would be recoded
BMI as Risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Body weight and height will be combined to report Body Mass Index in kg/m^2. Continuous variables are expressed as mean +/- standard deviation if they are normally distributed or as median and range otherwise. Independent Student's t-test is used for analyzing continuous variables with normal distribution and Mann-Whitney U test for continuous variables without normal distribution.
Age as Risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Age. Continuous variables are expressed as mean +/- standard deviation if they are normally distributed or as median and range otherwise. Independent Student's t-test is used for analyzing continuous variables with normal distribution and Mann-Whitney U test for continuous variables without normal distribution.
IIMs disease duration as Risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Disease duration in years. Continuous variables are expressed as mean +/- standard deviation if they are normally distributed or as median and range otherwise. Independent Student's t-test is used for analyzing continuous variables with normal distribution and Mann-Whitney U test for continuous variables without normal distribution.
Different subtypes of IIMs and risks for osteoporosis and osteopenia | at baseline
  Classification of IIMs according to Bohan and Peter criteria and presence of co-morbidities including chronic kidney disease, chronic liver disease, cardiovascular disease and diabetes mellitus. Personal history of previous vertebral or osteoporotic fracture and avascular necrosis. Chi-square test will be used to compare categorical variables.
Effect of medications on osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Drug history: Dosage of glucocorticoids (in milligram) at baseline and cumulative dose of glucocorticoids. Concomitant immunosuppressants and medication history.
Serum albumin level as risk factor in osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Serum albumin level
Serum C reactive protein level as risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Serum C reactive protein level
Erythrocyte sedimentation rate as risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Erythrocyte sedimentation rate
Serum creatine kinase as risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Serum Creatine kinase level
Disability as risk factor for osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  Health assessment questionnaire disability index at baseline
Effect of IIMS disease activity on osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  IIMs disease activity at baseline is measured by physician's and patient's global assessment by visual analogue scale
Effect of IIMs disease activity on osteoporosis and osteopenia in idiopathic inflammatory myopathies patients | at baseline
  IIMs disease activity at baseline is measured by manual muscle testing 8
New fractures during study period | during study period (12 months)
  New fractures including lumbar spine collapses during study period in two groups will be documented.
Adverse events associated with denosumab and zoledronic acid | throughout study period (12 months)
  Occurence of adverse events and early termination of denosumab and zoledronic acid would be documented. The following events will be monitored and documented:
  Mortality during treatment period Serious adverse events including infection requiring hopitalization, cardiac failure, stroke, myocardial infarction.
  Adverse events related to treatment: atypical femoral fracture, osteonecrosis of the jaw, back pain, arthralgia & mylagia, injection site reaction and allergy. Serious treatment related adverse events are adverse events leading to discontinuation of treatment. Related symptoms are documented during every clinic follow-up visits. All patient's medical and hospitalization record during the study period will also be reviewed by the investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- Kwong Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtis JR, Westfall AO, Allison J, Bijlsma JW, Freeman A, George V, Kovac SH, Spettell CM, Saag KG. Population-based assessment of adverse events associated with long-term glucocorticoid use. Arthritis Rheum. 2006 Jun 15;55(3):420-6. doi: 10.1002/art.21984. PMID 16739208
- [Background] Angeli A, Guglielmi G, Dovio A, Capelli G, de Feo D, Giannini S, Giorgino R, Moro L, Giustina A. High prevalence of asymptomatic vertebral fractures in post-menopausal women receiving chronic glucocorticoid therapy: a cross-sectional outpatient study. Bone. 2006 Aug;39(2):253-9. doi: 10.1016/j.bone.2006.02.005. Epub 2006 Mar 30. PMID 16574519
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (second of two parts). N Engl J Med. 1975 Feb 20;292(8):403-7. doi: 10.1056/NEJM197502202920807. No abstract available. PMID 1089199
- [Background] Isenberg DA, Allen E, Farewell V, Ehrenstein MR, Hanna MG, Lundberg IE, Oddis C, Pilkington C, Plotz P, Scott D, Vencovsky J, Cooper R, Rider L, Miller F; International Myositis and Clinical Studies Group (IMACS). International consensus outcome measures for patients with idiopathic inflammatory myopathies. Development and initial validation of myositis activity and damage indices in patients with adult onset disease. Rheumatology (Oxford). 2004 Jan;43(1):49-54. doi: 10.1093/rheumatology/keg427. Epub 2003 Jul 16. PMID 12867580
- [Background] Mok CC, Ying KY, To CH, Ho LY, Yu KL, Lee HK, Ma KM. Raloxifene for prevention of glucocorticoid-induced bone loss: a 12-month randomised double-blinded placebo-controlled trial. Ann Rheum Dis. 2011 May;70(5):778-84. doi: 10.1136/ard.2010.143453. Epub 2010 Dec 27. PMID 21187295
- [Background] Mok CC, Ho LY, Ma KM. Switching of oral bisphosphonates to denosumab in chronic glucocorticoid users: a 12-month randomized controlled trial. Bone. 2015 Jun;75:222-8. doi: 10.1016/j.bone.2015.03.002. Epub 2015 Mar 8. PMID 25761434
- [Background] Liu M, Guo L, Pei Y, Li N, Jin M, Ma L, Liu Y, Sun B, Li C. Efficacy of zoledronic acid in treatment of osteoporosis in men and women-a meta-analysis. Int J Clin Exp Med. 2015 Mar 15;8(3):3855-61. eCollection 2015. PMID 26064284
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Result] So H, Yip ML, Wong AK. Prevalence and associated factors of reduced bone mineral density in patients with idiopathic inflammatory myopathies. Int J Rheum Dis. 2016 May;19(5):521-8. doi: 10.1111/1756-185X.12405. Epub 2014 May 21. PMID 24848429
- [Result] Saag KG, Wagman RB, Geusens P, Adachi JD, Messina OD, Emkey R, Chapurlat R, Wang A, Pannacciulli N, Lems WF. Denosumab versus risedronate in glucocorticoid-induced osteoporosis: a multicentre, randomised, double-blind, active-controlled, double-dummy, non-inferiority study. Lancet Diabetes Endocrinol. 2018 Jun;6(6):445-454. doi: 10.1016/S2213-8587(18)30075-5. Epub 2018 Apr 6. PMID 29631782
- [Result] Reid DM, Devogelaer JP, Saag K, Roux C, Lau CS, Reginster JY, Papanastasiou P, Ferreira A, Hartl F, Fashola T, Mesenbrink P, Sambrook PN; HORIZON investigators. Zoledronic acid and risedronate in the prevention and treatment of glucocorticoid-induced osteoporosis (HORIZON): a multicentre, double-blind, double-dummy, randomised controlled trial. Lancet. 2009 Apr 11;373(9671):1253-63. doi: 10.1016/S0140-6736(09)60250-6. PMID 19362675